CLINICAL TRIAL: NCT03624270
Title: Risk-stratified Frontline Oral Arsenic Trioxide-based Induction in Newly Diagnosed Acute Promyelocytic Leukaemia
Brief Title: Oral Arsenic Trioxide for Newly Diagnosed Acute Promyelocytic Leukaemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL001
Record Dates: First submitted 2018-08-05; First posted 2018-08-10 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Acute Promyelocytic Leukemia
Keywords: Acute promyelocytic leukaemia; Oral arsenic trioxide
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Arsenic Trioxide; Tretinoin; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Frontline oral arsenic trioxide, ATRA and ascorbic acid (AAA) (Experimental): Induction:
  * Oral arsenic trioxide 10mg daily, all-trans retinoic acid (ATRA) (45mg/m2 per day in divided doses) and Ascorbic acid 1g daily for 42 days
  * Daunorubicin at 50mg/m2 daily for 3 days (omitted if WBC at diagnosis < 10 x 10^9/L; or age ≥ 65 years; or cardiac function impairment)
  * Hydroxyurea 2-4g per day if WBC > 5 x 10^9/L during the first 7 days of induction.
  Consolidation (for all patients):
  - Oral arsenic trioxide 10mg daily, all-trans retinoic acid (ATRA) (45mg/m2 per day in divided doses) and ascorbic acid 1g daily for 14 days every 28 days for 2 cycles
  Maintenance (for all patients):
  - Oral Arsenic trioxide 10mg daily, ATRA (45mg/m2 per day in divided doses) and ascorbic acid 1g daily for 2 weeks every 2 months for 24 months.
  Interventions: Drug: Oral arsenic Trioxide, ATRA and ascorbic acid

INTERVENTIONS:
Drug: Oral arsenic Trioxide, ATRA and ascorbic acid — Oral arsenic trioxide-based frontline induction, consolidation and maintenance will be provided to patients with newly diagnosed acute promyelocytic leukemia.

SUMMARY:
Acute promyelocytic leukemia (APL) is characterized by t(15;17)(q24;21) and the fusion gene PML-RARA. We have formulated an oral preparation of As2O3 (oral-As2O3), and shown that it is efficacious for APL in R1, inducing CR2 in more than 90% of patients. Furthermore, in an effort to prevent relapse, we have moved oral-As2O3 forward to the maintenance of CR1. This strategy results in favorable overall-survival (OS) and leukemia-free-survival (LFS), implying that prolonged treatment with oral-As2O3 may prevent relapses. Current protocols have incorporated i.v.-As2O3 in the treatment of newly-diagnosed APL. In regimens comprising i.v.-As2O3, ATRA and chemotherapy, 5-year overall survivals in excess of 90% is achieved. In this study, we evaluate the use of oral-As2O3 and ATRA based induction regimens in newly diagnosed patients with APL. In this study, we evaluate the efficacy and tolerability of frontline oral arsenic trioxide-based regimen in newly diagnosed patients with acute promyelocytic leukaemia

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients with acute promyelocytic leukaemia (APL) with t(15;17) (q24;q21)according to the World Health Organization (WHO) Classification 2016
* Patients aged ≥18 years
* Able and willing to comply with the study procedures and restrictions
* Having given voluntary written informed consent

Exclusion Criteria:

* ECOG performance status above 2
* Decompensated heart failure with left-ventricular ejection fraction of less than 40% and global hypokinesia on echocardiogram.
* Prolonged corrected QT interval (QTc) > 500ms, in the absence of electrolyte disturbances and medications known to prolong QTc
* Significant liver function derangement (Bilirubin > 3 times upper limit normal and/or ALT > 5 times upper limit of normal)
* Acute myeloid leukaemia with variant RARA translocation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival: Time (in months) from diagnosis to death or latest follow-up | 60 months
  Time (in months) from diagnosis to death (event) or latest follow-up (censor)
Leukemia-free survival: Time (in months) from first remission to relapse, death or latest follow-up | 60 months
  Time (in months) from first remission to relapse (event), death (event) or latest follow-up (censor)

SECONDARY OUTCOMES:
Treatment Toxicity Grade | 60 months
  Treatment toxicities by Eastern Cooperative Oncology (ECOG)-Common Toxicity Criteria (CTC)

CONTACTS AND LOCATIONS:
Overall Officials: Harinder Singh Harry Gill, MBBS, Principal Investigator — Department of Medicine, the University of Hong Kong
Locations (1):
- Department of Medicine, the University of Hong Kong, Queen Mary Hospital, Hong Kong, N/A = Not Applicable, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is no plan for IPD to be shared.